CLINICAL TRIAL: NCT03818984
Title: Safer Conception for HIV-infected Men Choosing to Conceive With At-risk Partners: Sinikithemba Kwabesilisa (Helping Men Have Healthy Babies)
Brief Title: Helping Men Have Healthy Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lynn T Matthews, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013P002693
Record Dates: First submitted 2018-12-07; First posted 2019-01-28 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: HIV/AIDS; HIV Prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Menogaril

STUDY DESIGN:
Intervention Model Description: Men will be offered 3 safer conception counseling sessions plus 2 booster sessions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Safer Conception Intervention (Experimental): Men will participate in 3 counseling sessions with a lay counselor. In the first session, the counselor will share information on the various safer conception strategies and help the participant think about developing a healthy plan. In the following 2 sessions, the counselor and the participant will work together to develop a healthy baby plan using motivational interviewing and problem solving. In the 2 booster sessions, the counselor and the participant will check in to evaluate the success of the plan and make changes as necessary.
  Interventions: Behavioral: Safer Conception for Men with At Risk Partners

INTERVENTIONS:
Behavioral: Safer Conception for Men with At Risk Partners — CBT based safer conception counseling with longitudinal follow-up and booster sessions. The primary outcome will be HIV RNA suppression at 6 months. Secondary outcomes include early ART uptake, adherence, serostatus disclosure, couples HIV counseling and testing uptake, and limiting unprotected sex to peak fertility.

SUMMARY:
Many men living with HIV (MLWH) want to have children. HIV-RNA suppression can minimize sexual HIV transmission risks while allowing for conception. The study will evaluate a safer conception intervention that leverages men's motivations to have healthy babies in order to promote serostatus disclosure and early ART initiation. The intervention is based on the investigators' Safer Conception Conceptual Framework, which considers individual, dyadic, and structural factors that affect periconception risk behavior.

DETAILED DESCRIPTION:
The study will evaluate and test a safer conception intervention that leverages men's motivations to have healthy babies in order to promote serostatus disclosure and early ART initiation. The intervention is based on a Safer Conception Conceptual Framework, which considers individual, dyadic, and structural factors that affect periconception risk behavior.

The researchers will conduct an open pilot to refine the intervention. The study will enroll men who want to have children with uninfected or unknown status female partners. Men will participate in three study sessions offering motivational interviewing and problem solving to help men develop a plan to have a healthy baby. The counseling will explore safer conception options including safe disclosure, delaying conception attempts until on ART with viral suppression, STI testing and treatment, timing condomless sex to peak fertility. The primary outcome is HIV RNA suppression at 12 weeks. Secondary outcomes include acceptability, feasibility, early ART uptake, adherence, serostatus disclosure, couples HIV counseling and testing uptake, and limiting unprotected sex to peak fertility.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as male
* Not on ART, or initiated ART within the past 3 months
* HIV-positive and status known for at least 1 (one) month,
* in care/patient at iThembalabantu clinic
* want to have a child in the next year,
* with a stable sexual pregnancy partner for at least 6 months,
* their pregnancy partner should be HIV-uninfected or HIV-status unknown,
* their pregnancy partner should not be known to be currently pregnant,
* have their own/ a mobile phone
* be fluent in either English or isiZulu and,
* able to participate in informed consent process
* not sterilized or known to be infertile

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
HIV RNA Suppression | 12 weeks
  Proportion of men achieving HIV-RNA suppression

SECONDARY OUTCOMES:
Uptake of ART | 12 weeks
  The proportion of men who initiate or continue ART
Uptake of HIV-serostatus disclosure | 12 weeks
  The proportion of men who report disclosure of HIV serostatus to pregnancy partner
Use of timing condomless sex to peak fertility | 12 weeks
  Through SMS surveys to assess weekly sexual behavior the study will evaluate the proportion of men who attempt to limit condomless sex to peak fertility

REFERENCES:
- [Derived] Matthews LT, Psaros C, Mathenjwa M, Mosery N, Greener LR, Khidir H, Hovey JR, Pratt MC, Harrison A, Bennett K, Bangsberg DR, Smit JA, Safren SA. Demonstration and Acceptability of a Safer Conception Intervention for Men With HIV in South Africa: Pilot Cohort Study. JMIR Form Res. 2022 May 4;6(5):e34262. doi: 10.2196/34262. PMID 35507406